CLINICAL TRIAL: NCT05243446
Title: Cardiorenal Effecs of Losartan in Kidney Transplant Recipients
Acronym: CELART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Collaborators: Medical University of Warsaw (Other); Pomeranian Medical University Szczecin (Other); Jagiellonian University (Other); Medical University of Bialystok (Other); Nicolaus Copernicus University (Other); Medical University of Silesia (Other); Poznan Regional Hospital (Unknown); Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Leszek Tylicki, Professor, Medical University of Gdansk
Other Study IDs: ST-4/CELART
Record Dates: First submitted 2022-01-24; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Renal Transplant Failure; Cardiovascular Complication
Keywords: angiotensin receptor blocker; kidney transplant recipients; albuminuria; cardiovascular disease; nephroprotection
MeSH Terms: conditions — Albuminuria; Cardiovascular Diseases | interventions — Losartan

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Study group: Hypotensive treatment including Losartan
  Interventions: Drug: Losartan
- Control group: Hypotensive treatment without renin-angiotensin-aldosteron system blockers.

INTERVENTIONS:
Drug: Losartan — losartan treatment
  Other Names: Lozap, Lorista, Xartan, Losacor
  Groups: Study group

SUMMARY:
The influence of Losartan to cardiovascular and renal outcomes in patients after renal transplatation.

DETAILED DESCRIPTION:
The benefits of cardio and nephroprotective properties of treatment with drugs blocking the renin angiotensin aldosterone system in the general population has already been shown. There are no data on the cardiac and renal effects of this type of treatment in patients after renal transplantation.

Therefore, the observational, case-control study was designed in a population of kidney transplant recipients.

The study group consists of patients treated with antihypertensive drugs including Losartan at a minimum dose of 50mg.

The control group consists of patients treated with antihypertensive drugs, without the renin angiotensin aldosterone system blockade.

Blood pressure will be controlled in accordance with the current recommendations.

The primary aim of this study is to determine whether, in renal transplant recipients with hypertension, losartan, angiotensin II receptor antagonist improves cardiovascular and graft outcome i.e. reduces incidence of cardiovascular complications and slows progression of graft insufficiency. Secondary objective is to determine whether losartan 1. delays the occurrence of cardiovascular complications, 2. slows progression of graft insufficiency, 3. is the safe drug in renal transplant recipients, 4. decrease albuminuria and other surrogate markers of graft injury or cardiovascular involvement.

ELIGIBILITY:
Inclusion Criteria:

740 patients, either sex, either non-diabetic or diabetic who underwent the kidney transplantation and who:

1. Are at least three months post-transplantation
2. Have hypertension.
3. Have an estimated glomerular filtration rate greater than or equal to 30 ml/min/1.73 m2

Exclusion Criteria:

1. Pregnant or the possibility of becoming so and breast feeding.
2. Angioedema from an Angiotensin Converting Enzyme (ACE) inhibitor or Angiotensin Receptor Blocker (ARB) in the history.
3. Serum potassium greater than 5.5 mmol/l on two or more occasions in the preceding three months.
4. Graft artery stenosis (i.e. psv of more than 200 cm/s in doppler usg)
5. Left ventricular dysfunction that requires an ACE inhibitor or an ARB
6. New immunosuppressive agent was started or previous immunosuppressant stopped in the three months prior to study entry or plan to switch immunosuppressive agents within next three months.
7. Currently on four or more blood pressure pills and have an average blood pressure over three visits greater than 150/100.
8. Currently on an ACE-inhibitor or an ARB or treatment with an ACE inhibitor or ARB after kidney transplantation lasted more than 3 months.
9. Had an acute coronary syndrome, episode of malignant hypertension, stroke or transient ischaemic attack in the three months prior to study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after renal transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 740 (Estimated)
Dates: Start 2015-09; Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of composite primary endpoint: | Up to 5 years
  Cardiovascular (CV) death and Resuscitated sudden death and Non-fatal myocardial infarction (MI) and Non-fatal stroke and Unplanned hospitalization for heart failure or unstable angina and Onset of end-stage renal disease (ESRD) and Doubling of baseline serum creatinine concentration, sustained for at least one month.

SECONDARY OUTCOMES:
Occurrence of cardiovascular complications | Up to 5 years
  Cardiovascular (CV) death and Resuscitated sudden death and Non-fatal myocardial infarction (MI) and Non-fatal stroke and Unplanned hospitalization for heart failure or unstable angina
Occurrence of renal complications | Up to 5 years
  ESRD or doubling of baseline serum creatinine
Decline in estimated glomerular filtration rate (eGFR) | Up to 5 years
  Difference in degree of eGFR reduction
Urine albumine concentration | after 6 months
  Difference in albuminuria in the measurements available for each patient
N-acetyl-β-D-glucosaminidase (NAG) urine excretion | after 6 months
  Difference in urine NAF in the measurements available for each patient
15-F2t-isoprostanes (isoprostanes) urine excretion | after 6 months
  differences in 15-F2t-isoprostanes (isoprostanes) urine excretion in the measurements available for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Leszek Tylicki, professor, Principal Investigator — Medical University of Gdansk
Locations (1):
- Medical University, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Undecided